CLINICAL TRIAL: NCT06994793
Title: Investigation of the Validity and Reliability of Gait and Jumping Parameters Measured With iSen Device in Healthy Adults
Brief Title: Validity and Reliability of Gait and Jump Parameters Measured by the iSen Device in Healthy Adults
Status: Recruiting | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Saniye Aydoğan Arslan, Associate Professor, Kırıkkale University
Other Study IDs: KirikkaleUni-iSenSağlıklı
Record Dates: First submitted 2025-05-06; First posted 2025-05-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-05

CONDITIONS: Healthy Adults; Gait Analysis; Jumping Performance; Reliability and Validity
Keywords: Gait Analysis; Jumping Performance; iSen Device; Wearable Sensors; Reliability; Validity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Adults: Healthy adult volunteers aged 18 to 35 years with no history of lower extremity surgery or any musculoskeletal, neurological, or systemic conditions that could affect gait or jumping performance. Participants were recruited from university departments and underwent gait and jumping assessments using the iSen and BTS G-Walk devices.

SUMMARY:
This study aims to evaluate the validity and reliability of gait and jumping parameters measured with the iSen device in healthy adults. Gait analysis is a valuable tool for assessing general health, cognitive performance, quality of life, and mortality. It is commonly used by clinicians to assess functional limitations resulting from neurological or orthopedic conditions and to guide treatment plans. Traditional gait assessments primarily focus on walking speed, but additional parameters such as step length, step time, and gait symmetry are crucial for a comprehensive analysis.

The study will also assess vertical jump performance, which is a surrogate measure of explosive lower limb strength and is commonly used in sports performance and injury prediction. The iSen device, a wearable and affordable sensor, will be compared to the validated BTS G-Walk system to evaluate the accuracy and consistency of its measurements. Participants aged 18-35 with no history of musculoskeletal, neurological, or systemic conditions will be included.

The study will be conducted at Gazi University and Kırıkkale University, where participants will undergo assessments of gait and jump performance using both iSen and BTS G-Walk devices. A test-retest reliability protocol will be employed with a seven-day interval between measurements. The results will provide evidence on the suitability of the iSen device for reliable and valid gait and jump measurements in clinical settings

DETAILED DESCRIPTION:
This study seeks to evaluate the validity and reliability of gait and jumping parameters measured with the iSen device in healthy adults. Gait analysis is an important tool in clinical settings as it provides valuable information about an individual's general health, cognitive performance, quality of life, and mortality risk. It is particularly useful for identifying functional limitations resulting from neurological or orthopedic conditions. Clinicians often rely on gait analysis to customize treatment plans, monitor individual progress, and assess the therapeutic benefits of interventions. Additionally, gait analysis can help identify underlying abnormalities and disorders that contribute to reduced functionality, thus aiding clinical decision-making.

Traditionally, clinical gait assessments focus on walking speed, typically measured using timed walking tests such as the 10-meter walk test or the 6-minute walk test. However, these assessments often fall short of providing a comprehensive evaluation, as they do not account for other important gait parameters such as step length, step time, or gait symmetry. Spatio-temporal gait parameters, such as walking speed, step time, step length, and step width, are essential for evaluating changes that may predict fall risk. Moreover, they are important for understanding motor function in a variety of populations.

Currently, laboratory-based equipment such as 3D motion capture systems and force plates are considered the gold standard for gait analysis due to their precision. However, these systems are often costly, require large spaces, and demand significant time for setup and analysis. As a result, they are not always accessible in clinical environments. In recent years, wearable accelerometers have gained popularity as an alternative for gait analysis. These devices offer several advantages, including low cost, portability, ease of use, and the ability to perform assessments in real-world settings, such as walking corridors. Notably, accelerometer-based gait analysis can be completed in a short period, typically within 10 minutes, making it an efficient option for clinical practice.

In addition to gait analysis, vertical jump performance is also a key parameter for assessing lower extremity strength and explosive power. Jumping performance can provide insights into athletic ability, physical fitness, and injury risk. Vertical jump height, in particular, is widely used by physiotherapists, trainers, and health professionals to assess strength, neuromuscular fatigue, and explosive power. Several methods are used to measure jump height, including contact mats, force plates, and accelerometers. However, force plates, considered the gold standard, are not portable and require specialized expertise to operate. As a result, wearable sensors like the iSen device have emerged as a practical and cost-effective alternative for jump performance analysis.

The iSen device is a wearable, wireless sensor that offers advantages over traditional laboratory-based equipment due to its portability, affordability, and ease of use. However, there is limited evidence regarding the validity and reliability of the iSen device in measuring gait and jump parameters. This study aims to fill this gap by comparing the iSen device with the validated BTS G-Walk system, which has demonstrated reliability and validity in gait and jump assessments. By evaluating the performance of the iSen device in measuring spatio-temporal gait parameters and jump performance, the study seeks to provide evidence for its potential clinical use.

The study will be conducted at Gazi University and Kırıkkale University, and will involve healthy adult participants aged 18-35 who meet the inclusion criteria. Participants will be screened for musculoskeletal, neurological, or systemic disorders that could affect their gait or jump performance. Each participant will undergo a series of assessments using both the iSen and BTS G-Walk devices. The assessments will include gait analysis in a 7-meter walking course, as well as vertical jump tests. To assess the test-retest reliability of the iSen device, participants will be re-assessed after a seven-day interval.

This study will contribute to the evidence base on the validity and reliability of the iSen device in measuring gait and jump parameters. The findings will provide valuable insights for clinicians and healthcare providers, helping them determine whether the iSen device can serve as a reliable, cost-effective alternative to traditional gait and jump assessment methods in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years. Voluntarily agree to participate in the study. No history of surgery in the lower extremities.

Exclusion Criteria:

* Any musculoskeletal, neurological, or systemic pathology that could affect gait or jumping performance.

Inability to comply with study procedures.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy adult volunteers aged 18 to 35 years who have not undergone lower extremity surgery and have no musculoskeletal, neurological, or systemic conditions that could affect gait or jumping performance. Participants will be recruited from Gazi University and Kırıkkale University, Department of Physiotherapy and Rehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Gait Speed | Baseline and 1 week later
  Gait speed (m/s) will be measured using the iSen system at baseline and one week later. At baseline, measurements will also be collected using the BTS G-Walk system for comparison to determine the validity of the iSen device in healthy adults.
Cadence | Baseline and 1 week later
  Cadence (steps/min) will be measured using the iSen system at baseline and one week later. At baseline, BTS G-Walk measurements will be used for validity comparison.
Step Length | Baseline and 1 week later
  Step length (m) will be measured using the iSen system at baseline and one week later. At baseline, BTS G-Walk measurements will be used for validity comparison.
Stance Phase Duration | Baseline and 1 week later
  Stance phase duration (%) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for validation.
Step Time | Baseline and 1 week later
  Step time (s) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for comparison.
Swing Phase Duration | Baseline and 1 week later
  Swing phase duration (%) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for validation.
Double Support Phase Duration | Baseline and 1 week later
  Double support phase duration (%) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for validation.
Single Support Phase Duration | Baseline and 1 week later
  Single support phase duration (%) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for validation
Pelvic Angles | Baseline and 1 week later
  Pelvic angles (degrees) will be measured using the iSen system at baseline and one week later. BTS G-Walk will be used at baseline for validation
Jump Height | Baseline and 1 week later
  Jump height (cm) will be measured during a countermovement jump using both the iSen and BTS G-Walk systems at baseline, and only the iSen system one week later. The highest value from three jumps will be recorded.
Take-off Force | Baseline and 1 week later
  Take-off force (kN) during a countermovement jump will be measured with the iSen and BTS G-Walk systems at baseline, and with iSen only one week later. The trial with the highest value will be analyzed.
Maximum Concentric Power | Baseline and 1 week later
  Maximum concentric power (kN) during a countermovement jump will be measured using both iSen and BTS G-Walk systems at baseline, and only iSen at one week. The value from the best trial will be used for analysis.
Landing Impact Force | Baseline and 1 week later
  Landing impact force (kN) will be assessed using both the iSen and BTS G-Walk systems at baseline, and the iSen system only at one-week follow-up.
Maximum Jump Velocity | Baseline and 1 week later
  Maximum vertical velocity (m/s) during a countermovement jump will be measured using the iSen and BTS G-Walk systems at baseline, and only iSen one week later. The maximum value from three trials will be recorded.
Take-off Velocity | Baseline and 1 week later
  Take-off velocity (m/s) will be assessed during a countermovement jump using both the iSen and BTS G-Walk systems at baseline, and only iSen at 1-week follow-up. The highest value will be selected.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirikkale University, Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Ridder R, Lebleu J, Willems T, De Blaiser C, Detrembleur C, Roosen P. Concurrent Validity of a Commercial Wireless Trunk Triaxial Accelerometer System for Gait Analysis. J Sport Rehabil. 2019 Aug 1;28(6):jsr.2018-0295. doi: 10.1123/jsr.2018-0295. PMID 30747572
- [Background] Yazici MV, Cobanoglu G, Yazici G. Test-retest reliability and minimal detectable change for measures of wearable gait analysis system (G-Walk) in children with cerebral palsy. Turk J Med Sci. 2022 Jun;52(3):658-666. doi: 10.55730/1300-0144.5358. Epub 2022 Jun 16. PMID 36326313